CLINICAL TRIAL: NCT02365961
Title: Reduction of Hip Arthroscopy Post-operative Pain Using Ultrasound-guided Fascia-iliaca Block
Brief Title: Hip Scope Fascia-iliaca (FI) Block Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Hawkins Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00038232
Record Dates: First submitted 2015-02-04; First posted 2015-02-19 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-02

CONDITIONS: Hip Dysplasia; Femoroacetabular Impingement; Acetabular Labrum Tear
Keywords: Hip Arthroscopy
MeSH Terms: conditions — Hip Dislocation; Femoracetabular Impingement | interventions — Clonidine; Epinephrine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FI Block (Experimental): Fascia iliaca block consisting of up to 60 mL of 0.35% ropivicaine at a dose of 3 mg/kg (with adjuvants of 100 mcg clonidine [per 60 mL] and epinephrine 1:400,000)
  Interventions: Drug: ropivicaine; Drug: clonidine; Drug: Epinephrine
- Local Injection (Active Comparator): Local anesthetic in the hip joint consisting of 30cc of 0.5% Noropin
  Interventions: Drug: Noropin

INTERVENTIONS:
Drug: ropivicaine
  Arms: FI Block
Drug: clonidine
  Arms: FI Block
Drug: Epinephrine
  Arms: FI Block
Drug: Noropin
  Arms: Local Injection

SUMMARY:
Patients undergoing a hip scope procedure will be recruited for this study. They will be randomized to either receive a nerve block or no nerve block (pain medicine only). Pain levels and clinical outcomes will be assessed through 3 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for outpatient hip arthroscopy
* American Society of Anesthesiologists (ASA) 1-3

Exclusion Criteria:

* Prior surgery on ipsilateral hip
* ASA 4-6
* Chronic narcotic usage over 6 months or more than the equivalent of 20mg of morphine per day
* Current or prior placement of a spinal cord stimulator or intrathecal pump for pain control purposes
* Allergy to amide local anesthetics
* Contraindication to regional anesthesia
* BMI > 40
* Females who are pregnant or plan to get pregnant during the course of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-04; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Kim, MD, Principal Investigator — Greenville Anesthesiology - Greenville Health System
Locations (1):
- Steadman Hawkins Clinic of the Carolinas - Greenville Health System, Greenville, South Carolina, United States

REFERENCES:
- [Derived] Glomset JL, Kim E, Tokish JM, Renfro SD, Seckel TB, Adams KJ, Folk J. Reduction of Postoperative Hip Arthroscopy Pain With an Ultrasound-Guided Fascia Iliaca Block: A Prospective Randomized Controlled Trial. Am J Sports Med. 2020 Mar;48(3):682-688. doi: 10.1177/0363546519898205. Epub 2020 Jan 30. PMID 31999469

RESULTS

PARTICIPANT FLOW:
Groups:
- FI Block: Fascia iliaca block consisting of up to 60 mL of 0.35% ropivicaine at a dose of 3 mg/kg (with adjuvants of 100 mcg clonidine [per 60 mL] and epinephrine 1:400,000)
  ropivicaine
  clonidine
  Epinephrine
- Local Injection: Local anesthetic in the hip joint consisting of 30cc of 0.5% Noropin
  Noropin
Period: Overall Study
Arm/Group | FI Block | Local Injection
Started | 41 | 43
Completed | 41 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FI Block | Local Injection | Total
Number analyzed (Participants) | 41 | 43 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 43 | 84
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 30 | 56
  Male | 15 | 13 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 40 | 40 | 80
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 37 | 37 | 74
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 41 | 43 | 84

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale
Description: Pain, as measured by Visual Analog Scale (VAS). Scores are ranged from 0-10, 0 is no pain and 10 is worst possible pain. The unit of measure is units on a scale.
Time Frame: 3 Months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | FI Block | Local Injection
Number analyzed (Participants) | 41 | 43
units on a scale | 2.65 [1.91 to 3.38] | 2.50 [1.77 to 3.23]

2. Secondary Outcome: Opioid Consumption
Description: Opioid consumption, as measured by narcotic usage (morphine milligram equivalents)
Time Frame: 3 Months
Measure: Mean (95% Confidence Interval); unit: morphine milligram equivalents
Arm/Group | FI Block | Local Injection
Number analyzed (Participants) | 41 | 43
morphine milligram equivalents | 26.87 [22.37 to 31.38] | 30.32 [26.03 to 34.61]

3. Other Pre Specified Outcome: Time in PACU
Description: Measured time subjects spent in the post anesthesia care unit.
Time Frame: Duration of PACU stay in minutes from end of surgery to discharge from PACA
Measure: Mean (95% Confidence Interval); unit: Minutes
Arm/Group | FI Block | Local Injection
Number analyzed (Participants) | 41 | 43
Minutes | 150.04 [128.95 to 171.20] | 151.59 [131.52 to 171.67]

4. Other Pre Specified Outcome: Total Number of Episodes of Nausea and Vomiting
Description: Occurrences of periods of nausea and vomiting
Time Frame: From end of surgery to discharge from PACU
Measure: Number; unit: Number of episodes
Arm/Group | FI Block | Local Injection
Number analyzed (Participants) | 41 | 43
Number of episodes | 11 | 7

5. Other Pre Specified Outcome: Hospital Readmission
Description: Number of participants that were readmitted to the hospital
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | FI Block | Local Injection
Number analyzed (Participants) | 41 | 43
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: Patients were assessed throughout their study participation, from surgery through the 3 month follow up.
Description: Both treatment are standard of care.
Arm/Group | FI Block | Local Injection
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/43
Other Adverse Events (participants affected / at risk) | 1/41 | 1/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FI Block (N=41) | Local Injection (N=43)
Hospital readmission (General disorders) | 1 (1) | 1 (1) — 2 patients were readmitted for postoperative pain control.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-29): https://cdn.clinicaltrials.gov/large-docs/61/NCT02365961/Prot_SAP_000.pdf